CLINICAL TRIAL: NCT01410227
Title: A Phase 3 Clinical Study to Determine the Pharmacokinetics, Safety and Efficacy of Recombinant Von Willebrand Factor : Recombinant Factor VIII (rVWF:rFVIII) and rVWF in the Treatment of Bleeding Episodes in Subjects Diagnosed With Von Willebrand Disease
Brief Title: Pharmacokinetics, Safety and Efficacy of Recombinant Von Willebrand Factor (rVWF) in the Treatment of Bleeding Episodes in Von Willebrand Disease (VWD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 071001; 2010-024108-84 (EudraCT Number)
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — Sodium Chloride; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PK 80 Arm (minimum of 22 subjects with severe VWD) (Experimental): PK assessment (80 IU/kg rVWF) + 12-month treatment period
  Interventions: Biological: Recombinant von Willebrand factor (rVWF); Biological: Recombinant factor VIIII (rFVIII)
- PK 50 Arm (14 subjects with type 3 VWD) (Experimental): Two single-blinded PK assessments (50 IU/kg rVWF + rFVIII/placebo) + 12-month treatment period
  Interventions: Biological: Recombinant von Willebrand factor (rVWF); Drug: Placebo; Biological: Recombinant factor VIIII (rFVIII)
- PK 50 Only Arm (minimum of 7 subjects with type 3 VWD) (Experimental): PK assessment (50 IU/kg rVWF) only, no treatment of bleeding episodes
  Interventions: Biological: Recombinant von Willebrand factor (rVWF); Drug: Placebo; Biological: Recombinant factor VIIII (rFVIII)
- Treatment Only (up to 7 subjects independent of VWD subtype) (Experimental): Treatment of bleeding episodes for a total of 12 months
  Interventions: Biological: Recombinant von Willebrand factor (rVWF); Biological: Recombinant factor VIIII (rFVIII)

INTERVENTIONS:
Biological: Recombinant von Willebrand factor (rVWF) — Intravenous administration
  Other Names: BAX 111; rVWF
Drug: Placebo — Syringe supplied with physiologic saline solution for infusion
  Other Names: saline; physiologic saline
  Arms: PK 50 Arm (14 subjects with type 3 VWD); PK 50 Only Arm (minimum of 7 subjects with type 3 VWD)
Biological: Recombinant factor VIIII (rFVIII) — Intravenous administration
  Other Names: rFVIII; ADVATE

SUMMARY:
The purpose of this Phase 3 study is to assess the pharmacokinetics of rVWF:rFVIII and rVWF, and to assess the safety and efficacy of rVWF:rFVIII and rVWF in the treatment of bleeding events in subjects with severe hereditary von Willebrand disease (VWD).

ELIGIBILITY:
Inclusion Criteria:

* Participant has been diagnosed with:

  1. Type 1 (Von Willebrand factor: Ristocetin cofactor activity (VWF:RCo) < 20 IU/dL) or,
  2. Type 2A (VWF:RCo < 20 IU/dL), Type 2B (as diagnosed by genotype), Type 2N (Factor VIII activity (FVIII:C) <10% and historically documented genetics), Type 2M or,
  3. Type 3 ( Von Willebrand factor antigen (VWF:Ag) ≤ 3 IU/dL) or,
  4. Severe Von Willebrand disease (VWD) with a history of requiring substitution therapy with von Willebrand factor concentrate to control bleeding
* Participant, who participates in the treatment for bleeding episodes, has had a minimum of 1 documented bleed (medical history) requiring VWF coagulation factor replacement therapy during the previous 12 months prior to enrollment.
* Participant has a Karnofsky score ≥ 60%
* Participant is at least 18 and not older than 65 years of age at enrollment
* If female of childbearing potential, participant presents with a negative pregnancy test
* Participant agrees to employ adequate birth control measures for the duration of the study
* Participant is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Participant has been diagnosed with pseudo VWD or another hereditary or acquired coagulation disorder other than VWD (eg qualitative and quantitative platelet disorders or elevated PT/international normalized ratio [INR] >1.4).
* Participant has a documented history of a VWF:RCo half-life of <6 hours.
* Participant has a history or presence of a VWF inhibitor at screening.
* Participant has a history or presence of a factor VIII (FVIII) inhibitor with a titer ≥0.4 BU (by Nijmegen assay) or ≥ 0.6 BU (by Bethesda assay).
* Participant has a known hypersensitivity to any of the components of the study drugs, such as mouse or hamster proteins.
* Participant has a medical history of immunological disorders, excluding seasonal allergic rhinitis/conjunctivitis, mild asthma, food allergies or animal allergies.
* Participant has a medical history of a thromboembolic event.
* Participant is HIV positive with an absolute CD4 count <200/mm3.
* Participant has been diagnosed with cardiovascular disease (New York Heart Association [NYHA] classes 1-4.
* Participant has an acute illness (eg, influenza, flu-like syndrome, allergic rhinitis/conjunctivitis, non-seasonal asthma) at screening.
* Participant has been diagnosed with significant liver disease as evidenced by any of the following: serum alanine aminotransferase (ALT) 5 times the upper limit of normal; hypoalbuminemia; portal vein hypertension (eg, presence of otherwise unexplained splenomegaly, history of esophageal varices).
* Participant has been diagnosed with renal disease, with a serum creatinine level ≥2 mg/dL.
* In the judgment of the investigator, the participant has another clinically significant concomitant disease (eg, uncontrolled hypertension) that may pose additional risks for the participant.
* Participant has been treated with an immunomodulatory drug, excluding topical treatment (eg, ointments, nasal sprays), within 30 days prior to enrollment
* Participant is pregnant or lactating at the time of enrollment.
* Participant has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an investigational product or investigational device during the course of this study.
* Participant has a history of drug or alcohol abuse within the 2 years prior to enrollment.
* Participant has a progressive fatal disease and/or life expectancy of less than 3 months.
* Participant is identified by the investigator as being unable or unwilling to cooperate with study procedures.
* Participant suffers from a mental condition rendering him/her unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude.
* Participant is in prison or compulsory detention by regulatory and/or juridical order

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (52):
- United States (10):
  - University of California Davis Cancer Center, Sacramento, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Illinois College of Medicine at Peoria, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Mary M Gooley Hemophilia Center and Rochester General Hospital, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Blood Center of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Perth Hospital, Perth, Western Australia
- Medical University Vienna, Vienna, Austria
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Bulgaria (2):
  - Specialized Haematological Hospital "Joan Pavel", Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
- University of Alberta Hospital, Edmonton, Alberta, Canada
- Germany (3):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Gerinnungszentrum Rhein-Ruhr, Duisburg
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz
- India (3):
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune
  - Sahyadri Speciality Hospital, Pune
  - Christian Medical College, Vellore
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Università degli Studi di Roma "La Sapienza", Roma
  - Ospedale San Bortolo, Vicenza
- Japan (3):
  - Nagoya University Hospital, Nagoya
  - Tokyo Medical University Hospital, Tokyo
  - Ogikubo Hospital, Tokyo
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
- Poland (4):
  - Hematology and Transplantology Clinic, University Clinic Centre - Medical University Hospital, Gdansk
  - Nicolaus Copernicus Provincial Specialist Hospital in Lodz Department of Hematology, Krakow
  - Institute of Haematology and Transfusion Medicine, Warsaw
  - Independent Public Clinical Hospital No. 1 in Wroclaw, Department of Hematology, blood cancer and Bone Marrow Transplantation, Wroclaw
- Russia (4):
  - Kirov Hematology and Blood Transfusion Research Institute under the Federal Medical and Biological Agency of Russia, Kirov
  - Territorial Clinical Hospital, Krasnoyarsk
  - Municipal Policlinic # 37, Saint Petersburg
  - Regional Pediatric Clinical Hospital #1, Yekaterinburg
- Spain (4):
  - Hospital Materno Infantil Teresa Herrera, A Coruña, Galicia
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Paz, Palma de Mallorca
  - Hospital Universitario Marques de Valdecilla, Santander
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skåne University Hospital (SUS), Malmo
- United Kingdom (4):
  - The Royal London Hospital, London
  - Royal Free Hospital, London
  - Hammersmith Hospital, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Gill JC, Castaman G, Windyga J, Kouides P, Ragni M, Leebeek FW, Obermann-Slupetzky O, Chapman M, Fritsch S, Pavlova BG, Presch I, Ewenstein B. Hemostatic efficacy, safety, and pharmacokinetics of a recombinant von Willebrand factor in severe von Willebrand disease. Blood. 2015 Oct 22;126(17):2038-46. doi: 10.1182/blood-2015-02-629873. Epub 2015 Aug 3. PMID 26239086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled (signed informed consent) from 30 sites in 15 countries.
Pre-assignment Details: 49 participants provided informed consent and were screened for the study, of which 37 were exposed to study product. Reasons for discontinuation were 6 screen failures, consent withdrawn by 3 participants, 1 physician decision, 1 participant received high doses of rFVIII for oral procedure and arm for which 1 participant was eligible was closed.
Groups:
- Arm 1: PK50 + Treatment: In Part A, (pharmacokinetic [PK] assessment followed by on-demand treatment for bleeding episodes [BEs] for 6 months) participants were initially infused either with 50 IU/kg recombinant von Willebrand Factor:von Willebrand Ristocetin cofactor (VWF:RCo rVWF) [rVWF] administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) [rVWF:rFVIII] or 50 IU/kg rVWF administered together with saline. Participants then crossed over to the alternate infusion after washout (PK). For on-demand treatment, participants received study product [VWF:rFVIII or rVWF], where BEs were initially treated with rVWF:rFVIII and subsequently with rVWF with or without rFVIII, based on FVIII levels (dose based on previous FVIII levels or if not available from the individual participant's PK data at discretion of investigator). In part, B participants continued to receive on-demand treatment for BEs with study product [VWF:rFVIII or rVWF] for a further 6 months.
- Arm 2: PK50 Only: In Part A, (pharmacokinetic [PK] assessment followed by on-demand treatment for bleeding episodes [BEs] for 6 months) participants were initially infused either with 50 IU/kg recombinant von Willebrand Factor:von Willebrand Ristocetin cofactor (VWF:RCo rVWF) [rVWF] administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) [rVWF:rFVIII] or 50 IU/kg rVWF administered together with saline. Participants then crossed over to the alternate infusion after washout (PK). For on-demand treatment, participants received study product [VWF:rFVIII or rVWF], where BEs were initially treated with rVWF:rFVIII and subsequently with rVWF with or without rFVIII, based on FVIII levels (dose based on previous FVIII levels or if not available from the individual participant's PK data at discretion of investigator). Participants then exited the study or could opt to sign informed consent to move to Arm 1 receive treatment for bleeding episodes with study product.
- Arm 3: PK80 + Treatment: In Part A, participants initially underwent a first PK assessment of an infusion of 80 IU/kg recombinant von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF]. After the first PK assessment participants received on demand treatment for bleeding episodes (BEs) with study product [VWF:rFVIII or rVWF], where BEs were initially treated with rVWF:rFVIII and subsequently with rWVF with or without rFVIII, based on FVIII levels. If FVIII levels not available, the individual participant's PK data was used to determine rFVIII dose at discretion of investigator. Participants received on-demand treatment for 6 months after the first study product infusion. After 6 months participants underwent a second PK assessment of an infusion of 80 IU/kg rVWF. In part B, participants continued to receive on-demand treatment for BEs with study product [VWF:rFVIII or rVWF] for a further 6 months.
- Arm 4: Treatment Only: In Part A, participants received on-demand treatment for bleeding episodes (BEs) with study product (recombinant von Willebrand Factor [rVWF] administered together with recombinant Factor VIII [rFVIII] (rVWF:rFVIII) or rVWF alone), where BEs were initially treated with rVWF:rFVIII and subsequently with rVWF with or without rFVIII, based on FVIII levels. If not available, the individual participant's PK data was used to determine rFVIII dose at discretion of investigator. Participants received on-demand treatment for 6 months after the first study product infusion. In part, B participants continued to receive on-demand treatment for BEs with study product [VWF:rFVIII or rVWF] for a further 6 months. No pharmacokinetic (PK) assessments were conducted in this arm.
Period: Overall Study
Arm/Group | Arm 1: PK50 + Treatment | Arm 2: PK50 Only | Arm 3: PK80 + Treatment | Arm 4: Treatment Only
Started | 8 | 8 | 15 | 6
Completed | 4 | 8 | 13 | 5
Not Completed | 4 | 0 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Met Excl. Criteria After Starting Study | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline consists of all participants in study [N=37] so is a total of the four arms described in Participant Flow (Arm 1: PK50 + Treatment [N=8]; Arm 2: PK50 Only [N=8]; Arm 3: PK80 + Treatment [N=15]; Arm 4: Treatment Only [N=6]).
Groups:
- All Subjects Treated With Study Product: All subjects treated with study product
Arm/Group | All Subjects Treated With Study Product
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: Years] | 37 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success for Treated Bleeding Episodes
Description: Treatment success was defined as the extent of control of bleeding episodes (BEs) using a mean efficacy rating score of <2.5 for a participant's BEs treated with study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) during the study period. Scores used: Excellent = 1 - actual infusions ≤ estimated number of infusions required to treat BE; no additional VWF required (all BEs); Good = 2 - >1-2 infusions (minor/moderate BEs) or <1.5 infusions (major BEs) greater than estimated required to control BE; no additional VWF required (all BEs); Moderate = 3 ≥ 3 infusions (minor/moderate BEs) or ≥ 1.5 infusions (major BEs) greater than estimated required to control BE; no additional VWF required (all BEs); None = 4 - severe uncontrolled bleeding or intensity of bleeding not changed; additional VWF required. Included participants with available primary efficacy rating (prospective-excluding gastrointestinal bleeds) in the Full Analysis Set.
Time Frame: For 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number (90% Confidence Interval); unit: Percent of participants
Groups:
- Full Analysis Set: Comprises of participants treated with study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) for whom at least one efficacy rating scale was available.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 18
Percent of participants | 100.0 [84.7 to 100.0]
Statistical Analysis 1: Comparison: Full Analysis Set; Test type: Non-Inferiority or Equivalence — The null hypothesis of the rate of subjects with a treatment success of <= 0.65 (H0: p <= 0.65) versus an alternative hypothesis of > 0.65 (HA: p > 0.65) was tested at the 5% one-sided level of significance. The proportion of subjects with treatment success under the alternative hypothesis was expected to be approximately 0.90. If 20 subjects were treated, the study provided 86% power to reject the null hypothesis; Clopper-Pearson; Clopper-Pearson = 100, 90% CI 2-sided [84.7 to 100]

2. Secondary Outcome: Percentage of Treated Bleeding Episodes With an Efficacy Rating of "Excellent" or "Good"
Description: Efficacy ratings "excellent" or "good" for the control of bleeding episodes (BEs) with study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) are defined as follows: Excellent - actual infusions ≤ estimated number of infusions required to treat BE; no additional von Willebrand Factor (VWF) required (all BEs); Good - >1-2 infusions (minor/moderate BEs) or <1.5 infusions (major BEs) greater than estimated required to control BE; no additional VWF required (all BEs). The data set included prospectively estimated BEs treated with study product with an available efficacy rating from participants in the Full Analysis Set
Time Frame: For 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number (90% Confidence Interval); unit: Percent of bleeding episodes
Units Other Than Participants: Bleeding episodes
Groups:
- Full Analysis Set: Comprised of participants treated with study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) for whom at least one efficacy rating scale was available.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 22
Number analyzed (Bleeding episodes) | 130
Percent of bleeding episodes | 100.0 [97.7 to 100.0]

3. Secondary Outcome: Percentage of Treated Bleeding Episodes With an Efficacy Rating of "Excellent" or "Good", Excluding Gastrointestinal Bleeds
Description: Efficacy ratings of "excellent" or "good" for the control of bleeding episodes (BEs) with study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) are defined as follows: Excellent - actual infusions ≤ estimated number of infusions required to treat BE; no additional von Willebrand Factor (VWF) required (all BEs); Good - >1-2 infusions (minor/moderate BEs) or <1.5 infusions (major BEs) greater than estimated required to control BE; no additional VWF required (all BEs). The data set included prospectively estimated BEs excluding gastrointestinal (GI) bleeds treated with study product with an available efficacy rating from participants in the Full Analysis Set.
Time Frame: For 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Geometric Mean (90% Confidence Interval); unit: Percent of bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 22
Number analyzed (Bleeding episodes) | 126
Percent of bleeding episodes | 100.0 [97.7 to 100.0]

4. Secondary Outcome: Number of Infusions of rVWF:rFVIII and/or rVWF Per Bleeding Episode
Description: The actual number of infusions of recombinant von Willebrand factor:recombinant factor VIII (rVWF:rFVIII) and/or rVWF required to treat a bleeding episode (BE). BEs were to be initially treated with an infusion of rVWF:rFVIII and subsequently with rVWF with or without rFVIII, based on FVIII levels, if available. In cases, where no FVIII levels were available, the individual participant's PK data was used to determine the rFVIII dose. The data set included prospectively estimated BEs treated with study product with an available efficacy rating from participants in the Full Analysis Set.
Time Frame: For 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Median (90% Confidence Interval); unit: Number of infusions
Units Other Than Participants: Bleeding episodes
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 22
Number analyzed (Bleeding episodes) | 192
Number of infusions | 1.0 [1.0 to 1.0]

5. Secondary Outcome: Number of Units of rVWF:rFVIII and/or rVWF Per Bleeding Episode
Description: The number of units is provided as the actual dose [IU/kg] of recombinant von Willebrand factor:recombinant factor VIII (rVWF:rFVIII) and/or rVWF required to treat a bleeding episode (BE). BEs were to be initially treated with an infusion of rVWF:rFVIII and subsequently with rVWF with or without rFVIII, based on FVIII levels, if available. In cases, where no FVIII levels were available, the individual participant's PK data was used to determine the rFVIII dose. The data set included prospectively estimated BEs treated with study product of known lot number with an available efficacy rating from participants in the Full Analysis Set.
Time Frame: For 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Median (90% Confidence Interval); unit: IU/kg
Units Other Than Participants: Bleeding episodes
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 22
Number analyzed (Bleeding episodes) | 174
IU/kg | 48.2 [43.9 to 50.2]

6. Secondary Outcome: Percentage of Participants Who Develop Inhibitory Antibodies to FVIII
Description: Development of neutralizing antibodies (inhibitors) to factor VIII (FVIII) was assessed by the Nijmegen modification of the Bethesda assay. Positive FVIII inhibitor tests were defined as ≥ 0.4 Bethesda units/mL (BU/mL) by the Nijmegen-modified Bethesda assay that is confirmed by a second test performed on an independent sample obtained 2-4 weeks following the first test. Category title includes number of participants [N] who provided data for the category.
Time Frame: For 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Percent of participants
Groups:
- Safety Analysis Set: Comprised of participants who were treated with study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) at least once during the study.
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Percent of participants
  Before 1st treatment with study product [N=37] | 0
  During 1st treatment until study end [N=27] | 0
  At final study visit [N=24] | 0

7. Secondary Outcome: Percentage of Participants Who Develop Inhibitory Antibodies to VWF
Description: Neutralizing antibodies (inhibitors) to Von Willebrand Factor Ristocetin cofactor (VWF:RCo), VWF collagen binding (VWF:CB) and VWF Factor VIII binding (VWF:FVIIIB) activities were measured using Nijmegen modification of the Bethesda assay. One Bethesda Unit (BU) is thereby defined as the amount of inhibitor that decreased the measured activity in the assays to 50% of that of the negative control samples. The assays were validated using human plasma samples from two type 3 VWD patients with low (1-2 BU/mL) and high (~10 BU/mL) titer inhibitors and plasma samples from non-human primates immunized with human rVWF (>100 BU/mL). Category title includes number of participants [N] who provided data for the category.
Time Frame: After signing informed consent until 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Percent of participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Percent of participants
  Before 1st treatment with study product [N=37] | 0
  During 1st treatment until study end [N=27] | 0
  At final study visit [N=24] | 0

8. Secondary Outcome: Percentage of Participants Who Develop Binding Antibodies to VWF
Description: The presence of total binding anti-VWF antibodies was determined by an enzyme-linked immunosorbent assay (ELISA) employing polyclonal anti-human immunoglobulin (Ig) antibodies (IgG, IgM and IgA). Category title includes number of participants [N] who provided data for the category.
Time Frame: After signing informed consent until 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Percent of participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Percent of participants
  Before 1st treatment with study product [N=37] | 0
  During 1st treatment until study end [N=28] | 0
  At final study visit [N=24] | 0

9. Secondary Outcome: Percentage of Participants Who Develop Binding Antibodies to CHO
Description: The presence of total binding anti-CHO antibodies was determined by measuring total immunoglobulin (Ig) antibodies (IgG, IgA, IgM) against Chinese Hamster Ovary (CHO) protein using an enzyme-linked immunosorbent assay (ELISA). Category title includes number of participants [N] who provided data for the category.
Time Frame: After signing informed consent until 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Percent of participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Percent of participants
  Before 1st treatment with study product [N=37] | 0
  During 1st treatment until study end [N=28] | 0
  At final study visit [N=24] | 0

10. Secondary Outcome: Percentage of Participants Who Develop Binding Antibodies to rFurin
Description: The presence of total binding anti-rFurin antibodies was determined by measuring total immunoglobulin (Ig) antibodies (IgG, IgA, IgM) against rFurin protein using an enzyme-linked immunosorbent assay (ELISA). Category title includes number of participants [N] who provided data for the category.
Time Frame: After signing informed consent until 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Percent of participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Percent of participants
  Before 1st treatment with study product [N=37] | 0
  During 1st treatment until study end [N=28] | 0
  At final study visit [N=24] | 0

11. Secondary Outcome: Percentage of Participants Who Develop Binding Antibodies to Mouse Immunoglobulin
Description: The presence of total binding anti-Murine immunoglobulin (IgG) antibodies was determined using an enzyme-linked immunosorbent assay (ELISA). Category title includes number of participants [N] who provided data for the category.
Time Frame: After signing informed consent until 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Percent of participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Percent of participants
  Before 1st treatment with study product [N=37] | 2.8
  During 1st treatment until study end [N=28] | 0
  At final study visit [N=24] | 0

12. Secondary Outcome: Percentage of Participants Who Had an Occurrence of Thrombotic Events
Time Frame: After signing informed consent until 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Percent of participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Percent of participants | 0

13. Secondary Outcome: Number of Adverse Events Related to Study Product Including Clinically Significant Changes in Laboratory Parameters and Vital Signs
Description: Adverse Events (AEs) related to study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) are described. Only laboratory parameters (hematology and clinical chemistry) and vital signs (physical examination, ECG) with clinically significant findings that are recorded as AEs are included. Categories presented as Severity-System Organ Class-Preferred Term Seriousness: serious adverse event (SAE); non serious adverse event (nsAE) System Organ Class: Cardiac disorders (CARD); General disorders and administration site conditions (GEN); Investigations (INV); Nervous system disorders (NERV); Skin and subcutaneous tissue disorders (SKN); Vascular disorders (VAS). Category title includes number of AEs [N] for the category.
Time Frame: For 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Number of Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Number analyzed (Adverse Events) | 125
Number of Adverse Events
  SAE-GEN-Chest discomfort [N=1] | 1
  SAE-INV-Heart rate increased [N=1] | 1
  nsAE-CARD-Tachycardia [N=1] | 1
  nsAE-GEN-Infusion site paraesthesia [N=1] | 1
  nsAE-INV-ECG T wave inversion [N=1] | 1
  nsAE-NERV-Dysgeusia [N=1] | 1
  nsAE-SKN-Pruritus generalized [N=1] | 1
  nsAE-VAS-Hot flush [N=1] | 1

14. Secondary Outcome: Number of Participants With Adverse Events Related to Study Product Including Clinically Significant Changes in Laboratory Parameters and Vital Signs
Description: Number of participants with Adverse Events (AEs) related to study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) are described. Only laboratory parameters (hematology and clinical chemistry) and vital signs (physical examination, ECG) with clinically significant findings that are recorded as AEs are included. Categories presented as Severity-System Organ Class-Preferred Term Seriousness: serious adverse event (SAE); non serious adverse event (nsAE) System Organ Class: Cardiac disorders (CARD); General disorders and administration site conditions (GEN); Investigations (INV); Nervous system disorders (NERV); Skin and subcutaneous tissue disorders (SKN); Vascular disorders (VAS).
Time Frame: For 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Number of participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Number of participants
  SAE-GEN-Chest discomfort | 1
  SAE-INV-Heart rate increased | 1
  nsAE-CARD-Tachycardia | 1
  nsAE-GEN-Infusion site paraesthesia | 1
  nsAE-INV-ECG T wave inversion | 1
  nsAE-NERV-Dysgeusia | 1
  nsAE-SKN-Pruritus generalized | 1
  nsAE-VAS-Hot flush | 1

15. Secondary Outcome: Number of Adverse Events by Infusion Related to Study Product Including Clinically Significant Changes in Laboratory Parameters and Vital Signs
Description: Adverse Events (AEs) by infusion related to study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) are described. Only laboratory parameters (hematology and clinical chemistry) and vital signs (physical examination, ECG) with clinically significant findings that are recorded as AEs are included. Categories presented as Severity-System Organ Class-Preferred Term Seriousness: serious adverse event (SAE); non serious adverse event (nsAE) System Organ Class: Cardiac disorders (CARD); General disorders and administration site conditions (GEN); Investigations (INV); Nervous system disorders (NERV); Skin and subcutaneous tissue disorders (SKN); Vascular disorders (VAS).
Time Frame: For 12 months after first infusion of rVWF:rFVIII or rVWF
Measure: Number; unit: Number of Adverse Events
Units Other Than Participants: Infusions
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 37
Number analyzed (Infusions) | 318
Number of Adverse Events
  SAE-GEN-Chest discomfort | 1
  SAE-INV-Heart rate increased | 1
  nsAE-CARD-Tachycardia | 1
  nsAE-GEN-Infusion site paraesthesia | 1
  nsAE-INV-ECG T wave inversion | 1
  nsAE-NERV-Dysgeusia | 1
  nsAE-SKN-Pruritus generalized | 1
  nsAE-VAS-Hot flush | 1

16. Secondary Outcome: PK50 - Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-∞/Dose) of VWF:RCo
Description: Area under the plasma concentration curve (AUC) from time 0 to infinity of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for subjects in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: PK evaluations at pre-infusion, then at 15, 30 and 60 mins, and 3, 6, 12, 24, 30, 48, 72 and 96 hrs post-infusion. PK evaluation timeframe for 28 ± 3 days after first infusion of study product which includes PK evaluation for both infusions and washout.
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Groups:
- PK50 Arms: Comprised of participants who underwent PK analysis of study product (50 IU/kg recombinant von Willebrand Factor (rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) [rVWF:rFVIII] or 50 IU/kg rVWF administered together with saline [rVWF]) i.e. a total of participants from Arm 1 [PK50+Treatment] and Arm 2 [PK50 only]. Participants in the PK50 arms have received at least one PK infusion and have provided data suitable for PK analysis. Only PK data included from the PK50 arms.
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
(hours*U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 32.4 [27.5 to 40.1]
  rVWF [N=14] | 32.7 [29.0 to 47.8]

17. Secondary Outcome: PK50 - Area Under the Plasma Concentration/Time Curve From Time 0 to 96 Hours (AUC0-96h/Dose) of VWF:RCo
Description: Area under the plasma concentration curve (AUC) from time 0 to 96 hours of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Groups:
- PK50 Arms: Comprised of participants who underwent PK analysis of study product (50 IU/kg recombinant von Willebrand Factor (rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) [rVWF:rFVIII] or 50 IU/kg rVWF administered together with saline [rVWF]) i.e. a total participants from Arm 1 [PK50+Treatment] and Arm 2 [PK50 only]. Participants in the PK50 arms have received at least one PK infusion and have provided data suitable for PK analysis. Only PK data included from the PK50 arms.
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
(hours*U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 31.6 [27.3 to 37.3]
  rVWF [N=14] | 31.3 [28.4 to 43.7]

18. Secondary Outcome: PK50 - Mean Residence Time of VWF:RCo
Description: Mean Residence Time (MRT) of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours
  rVWF:rFVIII [N=16] | 25.2 [20.0 to 30.1]
  rVWF [N=14] | 26.7 [22.7 to 36.0]

19. Secondary Outcome: PK50 - Clearance of VWF:RCo
Description: Clearance (CL) of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg/hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
dL/kg/hours
  rVWF:rFVIII [N=16] | 0.031 [0.025 to 0.041]
  rVWF [N=14] | 0.031 [0.021 to 0.035]

20. Secondary Outcome: PK50 - Incremental Recovery of VWF:RCo
Description: Incremental Recovery (IR) at the maximum plasma concentration of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (U/dL)/(U VWF: RCo/kg)
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
(U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 1.8 [1.6 to 2.4]
  rVWF [N=14] | 1.8 [1.5 to 2.2]

21. Secondary Outcome: PK50 - Elimination Phase Half-Life of VWF:Co
Description: Elimination Phase Half-Life (T1/2) of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant FVIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours
  rVWF:rFVIII [N=16] | 16.6 [14.7 to 20.4]
  rVWF [N=14] | 19.4 [15.5 to 31.3]

22. Secondary Outcome: PK50 - Volume of Distribution at Steady State of VWF:RCo
Description: Volume of Distribution at Steady State (Vss) of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
dL/kg
  rVWF:rFVIII [N=16] | 0.70 [0.66 to 0.93]
  rVWF [N=14] | 0.83 [0.70 to 0.97]

23. Secondary Outcome: PK50 - Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-∞/Dose) of VWF:Ag
Description: Area under the plasma concentration curve (AUC) from time 0 to infinity of von Willebrand Factor Antigen (VWF:Ag) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
(hours*U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 67.8 [55.1 to 81.7]
  rVWF [N=14] | 67.1 [55.6 to 80.5]

24. Secondary Outcome: PK50 - Area Under the Plasma Concentration/Time Curve From Time 0 to 96 Hours (AUC0-96h/Dose) of VWF:Ag
Description: Area under the plasma concentration curve (AUC) from time 0 to 96 hours of von Willebrand Factor Antigen (VWF:Ag) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
(hours*U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 62.1 [52.8 to 74.9]
  rVWF [N=14] | 62.2 [54.7 to 74.5]

25. Secondary Outcome: PK50 - Mean Residence Time of VWF:Ag
Description: Mean Residence Time (MRT) of von Willebrand Factor Antigen (VWF:Ag) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII] or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours
  rVWF:rFVIII [N=16] | 32.1 [29.8 to 41.1]
  rVWF [N=14] | 34.3 [30.4 to 41.4]

26. Secondary Outcome: PK50 - Clearance of VWF:Ag
Description: Clearance (CL) of von Willebrand Factor Antigen (VWF:Ag) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg/hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
dL/kg/hours
  rVWF:rFVIII [N=16] | 0.015 [0.013 to 0.018]
  rVWF [N=14] | 0.015 [0.013 to 0.018]

27. Secondary Outcome: PK50 - Incremental Recovery of VWF:Ag
Description: Incremental Recovery (IR) at the maximum plasma concentration of von Willebrand Factor Antigen (VWF:Ag) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (U/dL)/(U VWF: RCo/kg)
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
(U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 2.3 [2.0 to 2.5]
  rVWF [N=14] | 2.2 [1.9 to 2.5]

28. Secondary Outcome: PK50 - Elimination Phase Half-Life of VWF:Ag
Description: Elimination Phase Half-Life (T1/2) of von Willebrand Factor Antigen (VWF:Ag) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant FVIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours
  rVWF:rFVIII [N=16] | 21.8 [19.5 to 27.2]
  rVWF [N=14] | 25.2 [21.9 to 30.3]

29. Secondary Outcome: PK50 - Volume of Distribution at Steady State of VWF:Ag
Description: Volume of Distribution at Steady State (Vss) of von Willebrand Factor Antigen (VWF:Ag) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
dL/kg
  rVWF:rFVIII [N=16] | 0.50 [0.45 to 0.56]
  rVWF [N=14] | 0.49 [0.45 to 0.58]

30. Secondary Outcome: PK50 - Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-∞/Dose) of VWF:CB
Description: Area under the plasma concentration curve (AUC) from time 0 to infinity of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
(hours*U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 80.1 [68.4 to 95.0]
  rVWF [N=14] | 81.3 [71.2 to 99.8]

31. Secondary Outcome: PK50 - Area Under the Plasma Concentration/Time Curve From Time 0 to 96 Hours (AUC0-96h/Dose) of VWF:CB
Description: Area under the plasma concentration curve (AUC) from time 0 to 96 hours of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
(hours*U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 78.7 [66.5 to 90.5]
  rVWF [N=14] | 75.1 [69.2 to 97.0]

32. Secondary Outcome: PK50 - Mean Residence Time of VWF:CB
Description: Mean Residence Time (MRT) of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours
  rVWF:rFVIII [N=16] | 27.5 [22.7 to 32.1]
  rVWF [N=14] | 26.1 [25.1 to 33.2]

33. Secondary Outcome: PK50 - Clearance of VWF:CB
Description: Clearance (CL) of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg/hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
dL/kg/hours
  rVWF:rFVIII [N=16] | 0.012 [0.011 to 0.015]
  rVWF [N=14] | 0.012 [0.011 to 0.015]

34. Secondary Outcome: PK50 - Incremental Recovery of VWF:CB
Description: Incremental Recovery (IR) at the maximum plasma concentration of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (U/dL)/(U VWF: RCo/kg)
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
(U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 3.4 [3.0 to 3.7]
  rVWF [N=14] | 3.2 [2.8 to 3.7]

35. Secondary Outcome: PK50 - Elimination Phase Half-Life of VWF:CB
Description: Elimination Phase Half-Life (T1/2) of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant FVIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours
  rVWF:rFVIII [N=16] | 19.3 [14.9 to 23.4]
  rVWF [N=14] | 18.3 [17.4 to 24.8]

36. Secondary Outcome: PK50 - Volume of Distribution at Steady State of VWF:CB
Description: Volume of Distribution at Steady State (Vss) of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants[N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
dL/kg
  rVWF:rFVIII [N=16] | 0.35 [0.31 to 0.40]
  rVWF [N=14] | 0.36 [0.28 to 0.42]

37. Secondary Outcome: PK50 - Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-∞/Dose) of FVIII:C
Description: Area under the plasma concentration curve (AUC) from time 0 to infinity of Factor VIII activity (FVIII:C) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours*U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 145.4 [118.8 to 189.5]
  rVWF [N=14] | 113.0 [93.0 to 167.4]

38. Secondary Outcome: PK50 - Area Under the Plasma Concentration/Time Curve From Time 0 to 96 Hours (AUC0-96h/Dose) of FVIII:C
Description: Area under the plasma concentration curve (AUC) from time 0 to 96 hours of Factor VIII activity (FVIII:C) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII], or 50 IU/kg VWF:RCo rVWF administered together with saline (placebo) [rVWF] for participants in the PK50 arms (Arm 1 and Arm 2). Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours*U/dL)/(U VWF: RCo/kg)
  rVWF:rFVIII [N=16] | 127.8 [112.3 to 145.1]
  rVWF [N=14] | 101.8 [74.4 to 124.4]

39. Secondary Outcome: PK50 - Mean Residence Time of FVIII:C
Description: Mean Residence Time (MRT) of Factor VIII activity (FVIII:C) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII] for participants in the PK50 arms (Arm 1 and Arm 2).
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours | 44.0 [38.0 to 75.0]

40. Secondary Outcome: PK50 - Clearance of FVIII:C
Description: Clearance (CL) of Factor VIII activity (FVIII:C) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII] for participants in the PK50 arms (Arm 1 and Arm 2).
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg/hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
dL/kg/hours | 0.007 [0.006 to 0.009]

41. Secondary Outcome: PK50 - Incremental Recovery of FVIII:C
Description: Incremental Recovery (IR) at the maximum plasma concentration of Factor VIII activity (FVIII:C) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII] for participants in the PK50 arms (Arm 1 and Arm 2).
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (U/dL)/(U VWF: RCo/kg)
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 16
(U/dL)/(U VWF: RCo/kg) | 2.3 [1.9 to 2.7]

42. Secondary Outcome: PK50 - Elimination Phase Half-Life of FVIII:C
Description: Elimination Phase Half-Life (T1/2) of Factor VIII activity (FVIII:C) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant FVIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII] for participants in the PK50 arms (Arm 1 and Arm 2).
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
hours | 24.8 [20.1 to 50.5]

43. Secondary Outcome: PK50 - Volume of Distribution at Steady State of FVIII:C
Description: Volume of Distribution at Steady State (Vss) of Factor VIII activity (FVIII:C) after infusion of 50 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) administered together with 38.5 IU/kg recombinant Factor VIII (rFVIII) (ratio of 1.3:1±0.2) [rVWF:rFVIII] for participants in the PK50 arms (Arm 1 and Arm 2).
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg
Arm/Group | PK50 Arms
Number analyzed (Participants) | 16
dL/kg | 0.32 [0.29 to 0.44]

44. Secondary Outcome: PK80 - Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-∞/Dose) of VWF:RCo
Description: Area under the plasma concentration curve (AUC) from time 0 to infinity of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Groups:
- PK80 Arm: Comprised of participants who underwent PK analysis of study product (80 IU/kg recombinant von Willebrand Factor [rVWF]) i.e. participants from Arm 3 [PK80+Treatment]. Participants in this arm have received at least one PK infusion and have provided data suitable for PK analysis. Only PK data included in this arm.
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(hours*U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 36.9 [29.2 to 41.7]
  PK2 of rVWF [N=13] | 38.9 [28.1 to 43.3]

45. Secondary Outcome: PK80 - Area Under the Plasma Concentration/Time Curve From Time 0 to 96 Hours (AUC0-96h/Dose) of VWF:RCo
Description: Area under the plasma concentration curve (AUC) from time 0 to 96 hours of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(hours*U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 35.6 [28.9 to 41.2]
  PK2 of rVWF [N=13] | 37.9 [25.9 to 41.8]

46. Secondary Outcome: PK80 - Mean Residence Time of VWF:RCo
Description: Mean Residence Time (MRT) of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
hours
  PK1 of rVWF [N=15] | 26.4 [20.9 to 31.1]
  PK2 of rVWF [N=13] | 26.4 [23.7 to 32.8]

47. Secondary Outcome: PK80 - Clearance of VWF:RCo
Description: Clearance (CL) of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg/hours
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
dL/kg/hours
  PK1 of rVWF [N=15] | 0.027 [0.024 to 0.034]
  PK2 of rVWF [N=13] | 0.026 [0.023 to 0.036]

48. Secondary Outcome: PK80 - Incremental Recovery of VWF:RCo
Description: Incremental Recovery (IR) at the maximum plasma concentration Area under the plasma concentration curve (AUC) from time 0 to infinity of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 1.8 [1.7 to 2.2]
  PK2 of rVWF [N=13] | 1.8 [1.6 to 2.0]

49. Secondary Outcome: PK80 - Elimination Phase Half-Life of VWF:Co
Description: Elimination Phase Half-Life (T1/2) of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
hours
  PK1 of rVWF [N=15] | 18.4 [16.4 to 22.1]
  PK2 of rVWF [N=13] | 19.8 [15.2 to 23.6]

50. Secondary Outcome: PK80 - Volume of Distribution at Steady State of VWF:RCo
Description: Volume of Distribution at Steady State (Vss) of von Willebrand Factor Ristocetin cofactor (VWF:RCo) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study. PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
dL/kg
  PK1 of rVWF [N=15] | 0.78 [0.58 to 0.86]
  PK2 of rVWF [N=13] | 0.75 [0.58 to 1.01]

51. Secondary Outcome: PK80 - Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-∞/Dose) of VWF:Ag
Description: Area under the plasma concentration curve (AUC) from time 0 to infinity of von Willebrand Factor Antigen (VWF:Ag) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(hours*U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 66.6 [50.4 to 89.4]
  PK2 of rVWF [N=13] | 86.9 [54.9 to 100.5]

52. Secondary Outcome: PK80 - Area Under the Plasma Concentration/Time Curve From Time 0 to 96 Hours (AUC0-96h/Dose) of VWF:Ag
Description: Area under the plasma concentration curve (AUC) from time 0 to 96 hours of von Willebrand Factor Antigen (VWF:Ag) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(hours*U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 61.3 [48.8 to 73.7]
  PK2 of rVWF [N=13] | 77.4 [53.0 to 87.6]

53. Secondary Outcome: PK80 - Mean Residence Time of VWF:Ag
Description: Mean Residence Time (MRT) of von Willebrand Factor Antigen (VWF:Ag) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
hours
  PK1 of rVWF [N=15] | 38.4 [31.9 to 48.1]
  PK2 of rVWF [N=13] | 36.9 [30.0 to 50.8]

54. Secondary Outcome: PK80 - Clearance of VWF:Ag
Description: Clearance (CL) of von Willebrand Factor Antigen (VWF:Ag) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg/hours
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
dL/kg/hours
  PK1 of rVWF [N=15] | 0.015 [0.011 to 0.020]
  PK2 of rVWF [N=13] | 0.012 [0.010 to 0.018]

55. Secondary Outcome: PK80 - Incremental Recovery of VWF:Ag
Description: Incremental Recovery (IR) at the maximum plasma concentration Area under the plasma concentration curve (AUC) from time 0 to infinity of von Willebrand Factor Antigen (VWF:Ag) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 2.2 [1.9 to 2.6]
  PK2 of rVWF [N=13] | 2.4 [2.0 to 2.9]

56. Secondary Outcome: PK80 - Elimination Phase Half-Life of VWF:Ag
Description: Elimination Phase Half-Life (T1/2) of von Willebrand Factor Antigen (VWF:Ag) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
hours
  PK1 of rVWF [N=15] | 27.5 [22.5 to 34.0]
  PK2 of rVWF [N=13] | 24.8 [21.1 to 37.7]

57. Secondary Outcome: PK80 - Volume of Distribution at Steady State of VWF:Ag
Description: Volume of Distribution at Steady State (Vss) of von Willebrand Factor Antigen (VWF:Ag) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
dL/kg
  PK1 of rVWF [N=15] | 0.55 [0.46 to 0.61]
  PK2 of rVWF [N=13] | 0.50 [0.41 to 0.57]

58. Secondary Outcome: PK80 - Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-∞/Dose) of VWF:CB
Description: Area under the plasma concentration curve (AUC) from time 0 to infinity of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(hours*U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 73.9 [57.3 to 96.2]
  PK2 of rVWF [N=13] | 90.8 [66.0 to 105.2]

59. Secondary Outcome: PK80 - Area Under the Plasma Concentration/Time Curve From Time 0 to 96 Hours (AUC0-96h/Dose) of VWF:CB
Description: Area under the plasma concentration curve (AUC) from time 0 to 96 hours of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participatns from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(hours*U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 71.9 [57.0 to 89.8]
  PK2 of rVWF [N=13] | 88.1 [63.8 to 96.3]

60. Secondary Outcome: PK80 - Mean Residence Time of VWF:CB
Description: Mean Residence Time (MRT) of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
hours
  PK1 of rVWF [N=15] | 30.9 [24.3 to 35.0]
  PK2 of rVWF [N=13] | 28.7 [25.6 to 37.2]

61. Secondary Outcome: PK80 - Clearance of VWF:CB
Description: Clearance (CL) of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg/hours
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
dL/kg/hours
  PK1 of rVWF [N=15] | 0.014 [0.010 to 0.017]
  PK2 of rVWF [N=13] | 0.011 [0.010 to 0.015]

62. Secondary Outcome: PK80 - Incremental Recovery of VWF:CB
Description: Incremental Recovery (IR) at the maximum plasma concentration Area under the plasma concentration curve (AUC) from time 0 to infinity of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 3.1 [2.8 to 3.6]
  PK2 of rVWF [N=13] | 3.7 [2.7 to 4.0]

63. Secondary Outcome: PK80 - Elimination Phase Half-Life of VWF:CB
Description: Elimination Phase Half-Life (T1/2) of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
hours
  PK1 of rVWF [N=15] | 18.8 [16.6 to 24.9]
  PK2 of rVWF [N=13] | 20.9 [17.8 to 23.5]

64. Secondary Outcome: PK80 - Volume of Distribution at Steady State of VWF:CB
Description: Volume of Distribution at Steady State (Vss) of von Willebrand Factor Collagen Binding (VWF:CB) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: dL/kg
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
dL/kg
  PK1 of rVWF [N=15] | 0.39 [0.34 to 0.46]
  PK2 of rVWF [N=13] | 0.36 [0.33 to 0.40]

65. Secondary Outcome: PK80 - Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-∞/Dose) of FVIII:C
Description: Area under the plasma concentration curve (AUC) from time 0 to infinity of Factor VIII activity (FVIII:C) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(hours*U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 96.8 [64.0 to 126.5]
  PK2 of rVWF [N=13] | 94.8 [60.4 to 106.5]

66. Secondary Outcome: PK80 - Area Under the Plasma Concentration/Time Curve From Time 0 to 96 Hours (AUC0-96h/Dose) of FVIII:C
Description: Area under the plasma concentration curve (AUC) from time 0 to 96 hours of Factor VIII activity (FVIII:C) after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. Category title includes number of participants [N] who provided data for the category.
Time Frame: as for outcome 16
Measure: Median (95% Confidence Interval); unit: (hours*U/dL)/(U VWF: RCo/kg)
Arm/Group | PK80 Arm
Number analyzed (Participants) | 15
(hours*U/dL)/(U VWF: RCo/kg)
  PK1 of rVWF [N=15] | 81.7 [54.7 to 104.3]
  PK2 of rVWF [N=13] | 71.8 [49.6 to 89.2]

67. Secondary Outcome: PK80- Ratio of Intra-participant PK of VWF:RCo, VWF:Ag and VWF:CB at Baseline and After 6 Months
Description: Area under the plasma concentration curve (AUC) from time 0 to infinity per dose (AUC0-∞/dose) for von Willebrand Factor Ristocetin cofactor (VWF:RCo), von Willebrand Factor Antigen (VWF:Ag) and von Willebrand Factor Collagen Binding (VWF:CB). Each parameter was compared between the two PK assessments after infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] for participants in the PK80 arm (participants from Arm 3 with PK80 data only). PK assessment conducted at first infusion of 80 IU/kg rWVF [PK1] and the second infusion of 80 IU/kg rVWF after participants were treated on demand for bleeding episodes for at least 6 months since their first infusion of study product [PK2]. 13 participants had data available for this endpoint i.e. data for PK1 and PK2.
Time Frame: as for outcome 16
Population: Participants from the PK80 Arm who had pharmacokinetic (PK) data available after both the first infusion of 80 IU/kg recombinant von Willebrand Factor:von Willebrand Factor Ristocetin cofactor (VWF:RCo rVWF) [rVWF] [PK1] and the second infusion of 80 IU/kg rVWF [PK2].
Measure: Geometric Mean (90% Confidence Interval); unit: ratio of AUC0-∞/dose
Arm/Group | PK80 Arm
Number analyzed (Participants) | 13
ratio of AUC0-∞/dose
  AUC0-∞/dose - VWF:RCo | 0.9587 [0.8466 to 1.0857]
  AUC0-∞/dose - VWF:Ag | 1.0914 [1.0132 to 1.1757]
  AUC0-∞/dose - VWF:CB | 1.0666 [1.0004 to 1.1372]

ADVERSE EVENTS:
Time Frame: For 12 months after first infusion of recombinant von Willebrand Factor (rVWF) with or without recombinant Factor VIII (rVWF:rFVIII)
Groups:
- Safety Analysis Set: Comprises of participants who were treated with study product (recombinant von Willebrand Factor [rVWF] with or without recombinant factor VIII [rFVIII]) at least once during the study.
Arm/Group | Safety Analysis Set
Serious Adverse Events (participants affected / at risk) | 7/37
Other Adverse Events (participants affected / at risk) | 14/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=37)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Mesenteric haematoma (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Heart rate increased (Infections and infestations) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=37)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (4)
Vertigo (Ear and labyrinth disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4)
Infusion site paraesthesia (General disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Headache (Nervous system disorders) | 4 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or ≥12 months after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥40 days prior to submission or communication. Baxter may request an additional delay of ≤45 days eg, for intellectual property protection.